CLINICAL TRIAL: NCT04359810
Title: A Phase 2, Multi-Center, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Human Anti-SARS-CoV-2 Convalescent Plasma in Severely Ill Adults With COVID-19
Brief Title: Plasma Therapy of COVID-19 in Severely Ill Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Max O'Donnell (Other)
Collaborators: New York Blood Center (Other); Amazon, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Max O'Donnell, Florence Irving Associate Professor of Medicine and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS9924
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; COVID; Coronavirus; Convalescent plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: A total of 219 eligible subjects will be randomized in a 2:1 ratio to receive either convalescent plasma qualitatively positive for SARS-CoV-2 antibody (anti-SARS-CoV-2 plasma) or non-convalescent fresh frozen plasma (control plasma).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (anti-SARS-CoV-2 plasma) (Experimental): Convalescent plasma (1 unit; ~200-250 mL) collected from a volunteer who recovered from COVID-19 disease
  Interventions: Biological: Convalescent Plasma (anti-SARS-CoV-2 plasma)
- Non-convalescent Plasma (control plasma) (Active Comparator): Non-convalescent plasma (1 unit; ~200-250 mL) of standard plasma collected prior to December 2019
  Interventions: Biological: Non-convalescent Plasma (control plasma)

INTERVENTIONS:
Biological: Convalescent Plasma (anti-SARS-CoV-2 plasma) — Convalescent Plasma that contains antibody titers against SARS-CoV-2
  Arms: Convalescent Plasma (anti-SARS-CoV-2 plasma)
Biological: Non-convalescent Plasma (control plasma) — Non-convalescent plasma (does not contain antibody titers against SARS-CoV-2)
  Arms: Non-convalescent Plasma (control plasma)

SUMMARY:
This randomized blinded multi-center phase 2 trial will assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma among adults with severe COVID-19. Adults ≥18 years of age may participate. A total of 219 eligible subjects will be randomized in a 2:1 ratio to receive either high-titer anti-SARS-CoV-2 plasma or non-convalescent fresh frozen plasma (control plasma).

DETAILED DESCRIPTION:
There are few effective therapies for coronavirus disease 2019 (COVID-19) associated with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. Exposure to viruses results in an adaptive immune response that commonly include antibodies with neutralization activity. Plasma from subjects who have recovered from viral infections has been used to both prevent or treat disease. Notable examples of the successful use of convalescent plasma (CP) include influenza, measles, Argentine hemorrhagic fever, Middle East respiratory syndrome (MERS), Ebola and severe acute respiratory syndrome (SARS-CoV). Small clinical trials and observational studies of CP therapy in patients with COVID-19 have suggested a possible clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures or have a legally authorized representative available to do so.
* Age ≥18 years
* Evidence of SARS-CoV-2 infection by PCR test of naso-/oro-pharyngeal swab or tracheal aspirate sample within 14 days of randomization
* Peripheral capillary oxygen saturation (SpO2) ≤ 94% on room air or requiring supplemental oxygen, non-invasive or invasive mechanical ventilation at screening
* Evidence of infiltrates on chest radiography
* Females of childbearing age and males, must be willing to practice an effective contraceptive method or remain abstinent during the study period.

Exclusion Criteria:

* Participation in another clinical trial of anti-viral agent(s) for COVID-19
* Receipt of any anti-viral agent(s) with possible activity against SARS-CoV-2 <24 hours prior to study drug administration [1]
* Mechanically ventilated (including veno-venous (VV)-ECMO) ≥ 5 days
* Severe multi-organ failure
* History of prior reactions to transfusion blood products meeting definitive case definition criteria, at least severe severity, and probable or definite imputability per National Healthcare Safety Network (NHSN)/Centers for Disease Control and Prevention (CDC) criteria
* Known Immunoglobulin A (IgA) deficiency
* Females who are pregnant

  1. Use of remdesivir as treatment for COVID-19 is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max O'Donnell, MD, Principal Investigator — Columbia University
Locations (4):
- Columbia University Irving Medical Center/NYP, New York, New York, United States
- Brazil (3):
  - Hospital Federal dos Servidores do Estado, Rio de Janeiro
  - Hospital Geral de Nova Iguaçu, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Yes
The data-sharing plans for this study will be made available at a later date.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Austin PC, Fine JP. Practical recommendations for reporting Fine-Gray model analyses for competing risk data. Stat Med. 2017 Nov 30;36(27):4391-4400. doi: 10.1002/sim.7501. Epub 2017 Sep 15. PMID 28913837
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Li L, Zhang W, Hu Y, Tong X, Zheng S, Yang J, Kong Y, Ren L, Wei Q, Mei H, Hu C, Tao C, Yang R, Wang J, Yu Y, Guo Y, Wu X, Xu Z, Zeng L, Xiong N, Chen L, Wang J, Man N, Liu Y, Xu H, Deng E, Zhang X, Li C, Wang C, Su S, Zhang L, Wang J, Wu Y, Liu Z. Effect of Convalescent Plasma Therapy on Time to Clinical Improvement in Patients With Severe and Life-threatening COVID-19: A Randomized Clinical Trial. JAMA. 2020 Aug 4;324(5):460-470. doi: 10.1001/jama.2020.10044. PMID 32492084
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Liu STH, Lin HM, Baine I, Wajnberg A, Gumprecht JP, Rahman F, Rodriguez D, Tandon P, Bassily-Marcus A, Bander J, Sanky C, Dupper A, Zheng A, Nguyen FT, Amanat F, Stadlbauer D, Altman DR, Chen BK, Krammer F, Mendu DR, Firpo-Betancourt A, Levin MA, Bagiella E, Casadevall A, Cordon-Cardo C, Jhang JS, Arinsburg SA, Reich DL, Aberg JA, Bouvier NM. Convalescent plasma treatment of severe COVID-19: a propensity score-matched control study. Nat Med. 2020 Nov;26(11):1708-1713. doi: 10.1038/s41591-020-1088-9. Epub 2020 Sep 15. PMID 32934372
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] O'Donnell MR, Grinsztejn B, Cummings MJ, Justman JE, Lamb MR, Eckhardt CM, Philip NM, Cheung YK, Gupta V, Joao E, Pilotto JH, Diniz MP, Cardoso SW, Abrams D, Rajagopalan KN, Borden SE, Wolf A, Sidi LC, Vizzoni A, Veloso VG, Bitan ZC, Scotto DE, Meyer BJ, Jacobson SD, Kantor A, Mishra N, Chauhan LV, Stone EF, Dei Zotti F, La Carpia F, Hudson KE, Ferrara SA, Schwartz J, Stotler BA, Lin WW, Wontakal SN, Shaz B, Briese T, Hod EA, Spitalnik SL, Eisenberger A, Lipkin WI. A randomized double-blind controlled trial of convalescent plasma in adults with severe COVID-19. J Clin Invest. 2021 Jul 1;131(13):e150646. doi: 10.1172/JCI150646. PMID 33974559
- [Derived] Eckhardt CM, Cummings MJ, Rajagopalan KN, Borden S, Bitan ZC, Wolf A, Kantor A, Briese T, Meyer BJ, Jacobson SD, Scotto D, Mishra N, Philip NM, Stotler BA, Schwartz J, Shaz B, Spitalnik SL, Eisenberger A, Hod EA, Justman J, Cheung K, Lipkin WI, O'Donnell MR. Evaluating the efficacy and safety of human anti-SARS-CoV-2 convalescent plasma in severely ill adults with COVID-19: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Jun 8;21(1):499. doi: 10.1186/s13063-020-04422-y. PMID 32513308

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Started | 150 | 73
Completed | 150 | 73
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma) | Total
Number analyzed (Participants) | 150 | 73 | 223
Age, Customized [Count of Participants; unit: Participants]
  < 60 years old | 74 | 28 | 102
  60 - 69 years old | 35 | 24 | 59
  70 - 79 years old | 28 | 16 | 44
  >= 80 years old | 13 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 51 | 147
  Male | 54 | 22 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 24 | 73
  Brazil | 101 | 49 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Day 28 Severity Outcomes Using a 7-point Ordinal Scale of Clinical Status
Description: Compare the day 28 severity outcome amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups using a 7-point ordinal scale of clinical status. Seven-point ordinal scale for clinical assessment ranges from
  1 and 2: Not hospitalized 3: Hospitalized, not requiring supplemental oxygen 4: Hospitalized, requiring supplemental oxygen 5: Hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation 6: Hospitalized, requiring IMV, ECMO, or both 7: Dead Higher number means worse outcome
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 150 | 73
Participants
  Not hospitalized | 108 | 48
  Hospitalized, not requiring supplemental oxygen | 3 | 2
  Hospitalized, requiring supplemental oxygen | 7 | 1
  Hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation | 1 | 0
  Hospitalized, requiring IMV, ECMO, or both | 12 | 4
  Dead | 19 | 18

2. Secondary Outcome: Proportion of SARS-CoV-2 PCR Positivity
Description: Compare the proportion and duration of SARS-CoV-2 PCR positivity (via RT-PCR) amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups at days 0, 7, and 14.
Time Frame: Up to 14 days
Population: Data was not collected or analyzed.
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Levels of SARS-CoV-2 RNA
Description: Compare levels of SARS-CoV-2 RNA amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups at days 0, 7, and 14.
Time Frame: Up to 14 days
Population: Data was not collected or analyzed.
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Need for Supplemental Oxygen
Description: Compare duration of need for supplemental oxygen and/or mechanical ventilation amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 20 | 5
days | 6 [3 to 16] | 7 [3 to 11]

5. Secondary Outcome: Duration of Hospitalization
Description: Compare duration of hospitalization amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 23 | 7
days | 9 [6 to 28] | 8 [6 to 22]

6. Secondary Outcome: 28-day Mortality
Description: Compare up to 28-day mortality amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 150 | 73
Participants | 19 | 18

7. Secondary Outcome: Time-to-clinical Improvement In-hospital
Description: Compare time-to-clinical improvement in-hospital amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups, defined as the time to either an improvement of clinical status or alive discharge from the hospital, whichever comes first.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 150 | 73
days | 5 [4 to 6] | 7 [5 to 8]

8. Secondary Outcome: Host Genetic Differences at Day 0
Description: To assess for host genetic differences at Day 0 amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups.
Time Frame: Day 0
Population: Data was not collected or analyzed.
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Host Transcriptomic Differences at Days 0,7,14
Description: To assess for host transcriptomic differences at Day 0,7,14 amongst the anti-SARS-CoV-2 convalescent plasma and non-convalescent plasma groups.
Time Frame: Up to 14 days
Population: Data was not collected or analyzed.
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Adverse events and serious adverse events were monitored/assessed for a different population of participants (147 out of 150 Convalescent Plasma, and 72 out of 73 Non-convalescent Plasma).
  Adverse Events and serious adverse events were monitored/assessed without regard to the specific Adverse Event Term, given the circumstances surrounding the pandemic.
Arm/Group | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) | Non-convalescent Plasma (Control Plasma)
All-Cause Mortality (participants affected / at risk) | 19/150 | 18/73
Serious Adverse Events (participants affected / at risk) | 39/147 | 26/72
Other Adverse Events (participants affected / at risk) | 4/147 | 3/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) (N=147) | Non-convalescent Plasma (Control Plasma) (N=72)
Cardiovascular event (Vascular disorders) | 16 | 12
Pulmonary adverse event (Respiratory, thoracic and mediastinal disorders) | 24 | 16
Renal/metabolic adverse event (Renal and urinary disorders) | 7 | 5
Infectious adverse event (Infections and infestations) | 5 | 10
Hematologic adverse event (Blood and lymphatic system disorders) | 6 | 0
Inflammatory adverse event (Immune system disorders) | 1 | 0
Gastrointestinal/hepatic adverse event (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (Anti-SARS-CoV-2 Plasma) (N=147) | Non-convalescent Plasma (Control Plasma) (N=72)
Anemia, worsening (Blood and lymphatic system disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 0
Transfusion-related circulatory overload (Vascular disorders) | 2 | 1
Possible febrile non-hemolytic transfusion reaction (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04359810/Prot_SAP_000.pdf